CLINICAL TRIAL: NCT00486616
Title: Examination of Double-Lumen Tube Placement: Functional Electrical Impedance Tomography Versus Fibreoptic Bronchoscopy
Brief Title: Examination of Double-Lumen Tube Placement by Functional Electrical Impedance Tomography
Status: Completed | Type: Observational
Sponsor: University Hospital Freiburg (Other)
Other Study IDs: 117/07
Record Dates: First submitted 2007-06-13; First posted 2007-06-14 (Estimated); Last update posted 2008-02-18 (Estimated); Status verified 2007-08

CONDITIONS: Double-Lumen Tube Placement; One-Lung Ventilation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: electrical impedance tomography
Procedure: double-lumen tube placement

SUMMARY:
The purpose of this study is to determine whether functional electrical impedance tomography is suitable for examination of double-lumen tube placement compared with fibreoptic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* consent of the patient
* intubation with left- or right-sided double-lumen tube
* age >= 18 years

Exclusion Criteria:

* refusal by the patient
* contraindications for EIT-measurement (e.g. pacemaker, pregnancy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-05; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Steinmann, MD, Principal Investigator — Department of Anesthesia and Critical Care Medicine, University Hospital Freiburg
Locations (1):
- University Hospital Freiburg, Freiburg im Breisgau, Germany